CLINICAL TRIAL: NCT02750345
Title: A Three-Period Crossover Study to Determine the Bioequivalence of Two Oral Formulations Containing Nitisinone 10 mg Compared to Reference Formulation Orfadin In Healthy Subjects Under Fasting Conditions
Brief Title: Bioequivalence Study of Two Oral Nitisinone Formulations to Treat Hereditary Tyrosinemia (HT-1)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cycle Pharmaceuticals Ltd. (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CT-003; PXL227430 (Other: PAREXEL)
Record Dates: First submitted 2016-04-21; First posted 2016-04-25 (Estimated); Results first posted 2016-10-17 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Hereditary Tyrosinemia, Type I
Keywords: HT-1; Tyrosinemia; Nitisinone; Bioavailability; Healthy Volunteer; Food-Effect
MeSH Terms: conditions — Tyrosinemias | interventions — nitisinone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Sequence TP 1 - TP 2 - Reference (Experimental): Subjects will receive a single 10 mg tablet of Nitisinone (Test Product 1 (TP 1)) in treatment period 1, 10 mg tablet of Nitisinone Baked Tablet (Test Product 2 (TP 2)) in treatment period 2, and 10 mg hard capsule of Orfadin (Reference) in treatment period 3 under fasting conditions. Each treatment period will be separated by at least 23 calendar days of washout period.
  Interventions: Drug: Nitisinone; Drug: Nitisinone Baked Tablet; Drug: Orfadin
- Sequence TP 1 - Reference - TP 2 (Experimental): Subjects will receive a single 10 mg tablet of Nitisinone (Test Product 1) in treatment period 1, 10 mg hard capsule of Orfadin (Reference) in treatment period 2, and 10 mg tablet of Nitisinone Baked Tablet (Test Product 2) in treatment period 3 under fasting conditions. Each treatment period will be separated by at least 23 calendar days of washout period.
  Interventions: Drug: Nitisinone; Drug: Nitisinone Baked Tablet; Drug: Orfadin
- Sequence TP 2 - TP 1 - Reference (Experimental): Subjects will receive a single 10 mg tablet of Nitisinone Baked Tablet (Test Product 2) in treatment period 1, 10 mg tablet of Nitisinone (Test Product 1) in treatment period 2, and 10 mg hard capsule of Orfadin (Reference) in treatment period 3 under fasting conditions. Each treatment period will be separated by at least 23 calendar days of washout period.
  Interventions: Drug: Nitisinone; Drug: Nitisinone Baked Tablet; Drug: Orfadin
- Sequence TP 2 - Reference - TP 1 (Experimental): Subjects will receive a single 10 mg tablet of Nitisinone Baked Tablet (Test Product 2) in treatment period 1, 10 mg hard capsule of Orfadin (Reference) in treatment period 2, and 10 mg tablet of Nitisinone (Test Product 1) in treatment period 3, and under fasting conditions. Each treatment period will be separated by at least 23 calendar days of washout period.
  Interventions: Drug: Nitisinone; Drug: Nitisinone Baked Tablet; Drug: Orfadin
- Sequence Reference - TP 1 - TP 2 (Experimental): Subjects will receive a single 10 mg hard capsule of Orfadin (Reference) in treatment period 1, 10 mg tablet of Nitisinone (Test Product 1) in treatment period 2, and 10 mg tablet of Nitisinone Baked Tablet (Test Product 2) in treatment period 3 under fasting conditions. Each treatment period will be separated by at least 23 calendar days of washout period.
  Interventions: Drug: Nitisinone; Drug: Nitisinone Baked Tablet; Drug: Orfadin
- Sequence Reference - TP 2 - TP 1 (Experimental): Subjects will receive a single 10 mg hard capsule of Orfadin (Reference) in treatment period 1, 10 mg tablet of Nitisinone Baked Tablet (Test Product 2) in treatment period 2, and 10 mg tablet of Nitisinone (Test Product 1) in treatment period 3, and under fasting conditions. Each treatment period will be separated by at least 23 calendar days of washout period.
  Interventions: Drug: Nitisinone; Drug: Nitisinone Baked Tablet; Drug: Orfadin

INTERVENTIONS:
Drug: Nitisinone — A single oral dose of Nitisinone 10 mg Tablet will be administered.
Drug: Nitisinone Baked Tablet — A single oral dose of Nitisinone 10 mg Tablet (6 months @ 40°C/75% RH) will be administered.
  Other Names: Nitisinone (Baked)
Drug: Orfadin — A single oral dose of Orfadin 10 mg hard capsule will be administered.
  Other Names: Nitisinone

SUMMARY:
The purpose of this study is to determine whether Nitisinone 10 mg Tablets (Test Product 1) and Nitisinone 10 mg Tablets 'Baked' for 6 months @ 40°C/75% RH (Test Product 2) are bioequivalent to the reference product Orfadin 10 mg hard capsules.

DETAILED DESCRIPTION:
The specific aim is to conduct a randomized, single dose, three-period crossover bioequivalence study in at least 18 healthy male and female subjects at a single study center to evaluate the in vivo performance of two formulations of Nitisinone 10 mg and the reference product Orfadin under fasting.

A total of 24 healthy female and male volunteers (age 18 to 55 years old) will be entered into the study. Volunteers will be determined to be free of significant medical conditions as assessed by medical history, physical examination, and blood and urine tests. Volunteers will be randomly allocated to a treatment sequence, before administration of investigational medicinal product (IMP) under fasting conditions.

There will be a minimum 23 calendar days washout between treatments. Blood samples will be collected at pre-dose (0 hours) and at 15 minutes, 30 minutes, 1 hour, 2 hours, 2 hours and 30 minutes, 3 hours, 3 hours and 30 minutes, 4 hours, 5 hours, 6 hours, 7 hours, 8 hours, 10 hours, 12 hours, 24 hours, 36 hours, 48 hours, 72 hours, 96 hours and 120 hours post-dose (total: 21 samples per treatment period).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects, 18 to 55 years (both inclusive) at signing of informed consent.
* Body Mass Index (BMI) between 18.5 and 30 kg/m2 (inclusive).
* Body mass not less than 50 kg.
* Medical history, vital signs, physical examination, standard 12-lead electrocardiogram (ECG) and laboratory investigations must be clinically acceptable or within laboratory reference ranges for the relevant laboratory tests, unless the investigator considers the deviation to be irrelevant for the purpose of the study.
* Non-smokers.
* Females, if:

Of childbearing potential, the following conditions are to be met:

* Negative pregnancy test If this test is positive, the subject will be excluded from the study. In the rare circumstance that a pregnancy is discovered after the subject received IMP, every attempt must be made to follow her to term.
* Not lactating
* Abstaining from sexual activity (if this is the usual lifestyle of the subject) or must agree to use an accepted method of contraception, and agree to continue with the same method throughout the study Examples of reliable methods of contraception include non-hormonal intrauterine device, and barrier methods combined with an additional contraceptive method. In this study the concomitant use of hormonal contraceptives is NOT allowed. Other methods, if considered by the investigator as reliable, will be accepted.
* Written consent given for participation in the study.

Exclusion Criteria:

* Evidence of psychiatric disorder, antagonistic personality, poor motivation, emotional or intellectual problems likely to limit the validity of consent to participate in the study or limit the ability to comply with protocol requirements.
* Current alcohol use > 21 units of alcohol per week for males and > 14 units of alcohol per week for females.
* Consumption of more than 5 cups of coffee (or equivalent amounts of caffeine) per day.
* Regular exposure to substances of abuse (other than alcohol) within the past year.
* Use of any medication, prescribed or over-the-counter or herbal remedies, within 2 weeks before the first administration of IMP except if this will not affect the outcome of the study in the opinion of the investigator.

In this study the concomitant use of hormonal contraceptives is NOT allowed.

* Participation in another study with an experimental drug, where the last administration of the previous IMP was within 8 weeks (or within 10 elimination half-lives for chemical entities or 2 elimination half-lives for antibodies or insulin), whichever is the longer) before administration of IMP in this study, at the discretion of the investigator.
* Treatment within the previous 3 months before the first administration of IMP with any drug with a well-defined potential for adversely affecting a major organ or system.
* A major illness during the 3 months before commencement of the screening period.
* History of hypersensitivity or allergy to the IMP or its excipients or any related medication.
* History of bronchial asthma or any other bronchospastic disease.
* History of convulsions.
* History of porphyria.
* Relevant history or laboratory or clinical findings indicative of acute or chronic disease, likely to influence study outcome.
* Donation or loss of blood equal to or exceeding 500 mL during the 8 weeks before the first administration of IMP.
* Diagnosis of hypotension made during the screening period.
* Diagnosis of hypertension made during the screening period or current diagnosis of hypertension.
* Resting pulse of > 100 beats per minute or < 40 beats per minute during the screening period, either supine or standing.
* Positive testing for human immunodeficiency virus (HIV), Hepatitis B and Hepatitis C.
* Positive urine screen for drugs of abuse. In case of a positive result the urine screen for drugs of abuse may be repeated once at the discretion of the investigator.
* Positive urine screen for tobacco use.
* Positive pregnancy test.
* Female subjects that are pregnant or breastfeeding.
* Difficulty in swallowing.
* Any specific investigational product safety concern.
* Vulnerable subjects, e.g. persons in detention.
* Subjects with current keratopathy, or other clinically significant abnormalities found by slit-lamp examination (cataracts) at the discretion of the investigator.
* Concomitant use of medications that are metabolized by CYP2C9 (ibuprofen, diclofenac and indomethacin).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: André Nell, Principal Investigator — +27 51 410 3046
Locations (1):
- Bloemfontein Early Phase Clinical Unit, PAREXEL International (South Africa), Bloemfontein, Free State, South Africa

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Intervention 1
Arm/Group | Sequence TP 1 - TP 2 - Reference | Sequence TP 1 - Reference - TP 2 | Sequence TP 2 - TP 1 - Reference | Sequence TP 2 - Reference - TP 1 | Sequence Reference - TP 1 - TP 2 | Sequence Reference - TP 2 - TP 1
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0
Period: Intervention 2
Arm/Group | Sequence TP 1 - TP 2 - Reference | Sequence TP 1 - Reference - TP 2 | Sequence TP 2 - TP 1 - Reference | Sequence TP 2 - Reference - TP 1 | Sequence Reference - TP 1 - TP 2 | Sequence Reference - TP 2 - TP 1
Started | 4 | 4 | 4 | 4 | 3 | 4
Completed | 4 | 4 | 4 | 4 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Intervention 3
Arm/Group | Sequence TP 1 - TP 2 - Reference | Sequence TP 1 - Reference - TP 2 | Sequence TP 2 - TP 1 - Reference | Sequence TP 2 - Reference - TP 1 | Sequence Reference - TP 1 - TP 2 | Sequence Reference - TP 2 - TP 1
Started | 4 | 4 | 4 | 4 | 3 | 4
Completed | 4 | 4 | 4 | 4 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Grouped by all participants as this is how overall data has been collected.
Arm/Group | All Study Participants
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 21
Race/Ethnicity, Customized [Number; unit: Participants]
  Black | 16
  Caucasian | 7
  Mixed Race | 1
Region of Enrollment [Number; unit: participants]
  South Africa | 24

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: 0 - 120 hours post-dose
Population: All subjects for whom the primary pk parameters Cmax and AUC (0-120) could be calculated for at least two treatment periods (where one of which is the reference product), and who had no major protocol deviations thought to impact on the analysis of pk data were included in the statistical pk analysis for the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Test Product 1: 10 mg Nitisinone Tablet
- Test Product 2: Nitisinone 10 mg Tablet (6 months @ 40°C/75% RH)
- Reference Product: ORFADIN®, 10 mg hard capsule
Arm/Group | Test Product 1 | Test Product 2 | Reference Product
Number analyzed (Participants) | 23 | 23 | 23
ng/mL | 1277.77 (17.8) | 1272.34 (16.6) | 1339.79 (17.3)

2. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC(0-120))
Time Frame: 0 - 120 hours post-dose
Population: All subjects for whom the primary Pk parameters Cmax and AUC (0-120) could be calculated for at least 2 treatment periods (where one of the treatment includes the reference product), and who had no major protocol deviations thought to impact the analysis of the pk data were included for the statistical pk analysis for the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Groups:
- Treatment Period 1: 10 mg Nitisinone Tablet
- Treatment Period 2: Nitisinone 10 mg Tablet (6 months @ 40°C/75% RH)
Arm/Group | Treatment Period 1 | Treatment Period 2 | Reference Product
Number analyzed (Participants) | 23 | 23 | 23
hr*ng/mL | 77874.13 (19.3) | 77295.02 (20.00) | 78672.56 (17.4)

3. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC(0-72))
Time Frame: 0 - 72 hours post-dose
Population: All subjects for whom the primary pk parameters Cmax and AUC (0-120) could be calculated for at least 2 treatment periods (where one of the treatment periods must be the reference product), and who had no major protocol deviations thought to impact on the analysis of the pk data were included in the statistical pk analysis for the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Treatment Period 1 | Treatment Period 2 | Reference Product
Number analyzed (Participants) | 23 | 23 | 23
hr*ng/mL | 57838.41 (20.0) | 57497.79 (18.7) | 59013.52 (15.7)

4. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve, With Extrapolation to Infinity (AUC(0-∞))
Time Frame: 0 - 120 hours post-dose
Population: All subjects for whom the primary pk parameters Cmax and AUC (0-120) could be calculated for at least 2 treatment periods (where one of which is the reference product), and who had no major protocol deviations thought to impact on the analysis of pk data were included in the statistical pk analysis for the study
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Treatment Period 1 | Treatment Period 2 | Reference Product
Number analyzed (Participants) | 23 | 23 | 23
hr*ng/mL | 104495.96 (26.6) | 105117.79 (25.4) | 106892.31 (23.9)

5. Secondary Outcome: Time to Maximum Observed Plasma Concentration (Tmax)
Time Frame: 0 - 120 hours post-dose
Population: All subjects for whom the primary pk parameters Cmax and AUC (0-120) could be calculated for at least 2 treatment periods (where one of which must be the reference product), and who had no major protocol deviations thought to impact on the analysis of pk data were included in the statistical analysis for the study.
Measure: Median (Full Range); unit: hr
Arm/Group | Treatment Period 1 | Treatment Period 2 | Reference Product
Number analyzed (Participants) | 23 | 23 | 23
hr | 3.5 [1 to 4] | 4.0 [2 to 10] | 2.5 [0.5 to 10]

6. Secondary Outcome: Terminal Elimination Rate Constant (λz)
Time Frame: 0 - 120 hours post-dose
Population: All subjects for whom the primary pk parameters Cmax and AUC (0-120) could be calculated for at least 2 treatment periods (where one of which must be the reference product), and who had no major protocol deviations thought to impact on the analysis of pk data were included in the statistical pk analysis for the study
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hr
Arm/Group | Treatment Period 1 | Treatment Period 2 | Reference Product
Number analyzed (Participants) | 23 | 23 | 23
1/hr | 0.012 (15.8) | 0.011 (20.1) | 0.012 (21.1)

7. Secondary Outcome: Apparent Terminal Elimination Half-life (t1/2)
Time Frame: 0 - 120 hours post-dose
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Treatment Period 1 | Treatment Period 2 | Reference Product
Number analyzed (Participants) | 23 | 23 | 23
hr | 58.668 (15.8) | 60.780 (20.1) | 59.904 (21.1)

ADVERSE EVENTS:
Arm/Group | Test Product 1 | Test Product 2 | Reference Product
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23 | 0/24
Other Adverse Events (participants affected / at risk) | 3/23 | 1/23 | 1/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test Product 1 (N=23) | Test Product 2 (N=23) | Reference Product (N=24)
Flu (Infections and infestations) | 0 | 1 | 0
Vomit (Gastrointestinal disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0
Cold (Infections and infestations) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No